CLINICAL TRIAL: NCT04448145
Title: Characterizing SARS-CoV-2 Persistence in Host Reservoirs, Post-viral Sequelae, and Associations With Host and Viral Determinants in a Cohort of Convalescent COVID-19 Cases
Brief Title: Determinants of SARS (Severe Acute Respiratory Syndrome)-COV2 (COVID-19) Persistence After Convalescence
Acronym: C-PIC
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAS9722
Record Dates: First submitted 2020-06-24; First posted 2020-06-25 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: COVID-19; Corona Virus Infection; SARS-CoV 2
Keywords: Novel Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, Nasal Swab, Blood, Stool, Semen, Breastmilk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Positive: Participants who have been diagnosed with COVID-19 or experienced symptoms of COVID-19.
- COVID-19 Negative: Participants who have never tested positive for COVID-19.

SUMMARY:
The 2019-2020 COVID-19 pandemic is the largest outbreak in recent history. It is not known how long after someone gets sick with COVID-19 and recovers that they can still infect other people. It is also not known how quickly people make antibodies against the virus, which help clear infection from the body. The investigators will enroll 300 people who had COVID-19 based on lab testing or confirmed exposure to participate. An additional 25 participants who have never tested positive for COVID and have not had the vaccine will be enrolled as negative controls. Participants will complete a survey at enrollment. The investigators will also collect blood, nose swab, saliva, stool, semen, and breast milk to test for the virus. The investigators will ask participants to complete a survey and give specimens up to 12 times over 24 months. This information will be used to study how long the virus can live in different parts of the body, antibody development, and post-infectious complications. The investigators hope that this information will allow medical and public health providers to make recommendations to better care for patients in the convalescent phase of COVID-19 infection.

DETAILED DESCRIPTION:
This is an observational prospective cohort study of confirmed cases of COVID-19 recruited from communities surrounding New York City. 325 participants will be recruited from NewYork-Presbyterian (NYP)-Columbia hospital, the community using flyers and snowball sampling, and by contacting participants who are already participating in a Columbia University Irving Medical Center (CUIMC) COVID-19 related study and have given consent to be contacted about participation in related research studies. Candidates will be eligible to participate if they have received a laboratory confirmed diagnosis of COVID-19 or were symptomatic and had a known contact with a confirmed case of COVID-19, and are over the age of 7. Participants who were diagnosed empirically due to symptoms and exposure yet test negative by Reverse transcription polymerase chain reaction (RT-PCR) and serology at baseline will not be considered infected with SARS-CoV-2 and may be excluded. Participants will be consented prior to participation in any study activities and will be prospectively followed for 96 weeks. At baseline, an enrollment survey will be administered that includes demographics, comorbidities, and characteristics of their COVID-19 illness (e.g., exposure, symptom onset, symptom duration, severity of symptoms) and will provide blood and host reservoir site samples. Participants will be followed for a 24 month period after symptom onset, with a maximum of 12 visits.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed SARS-CoV-2 using currently available laboratory testing techniques (e.g.,RT-PCR, Immunoglobulin M (IgM) /IgG) or clinical history compatible with a COVID-19 like illness(fever, cough, shortness of breath).
* Negative participants with no known prior COVID-19 diagnosis or COVID vaccine
* At least 7 years of age
* Participants are eligible to provide semen and breast milk samples if they are 18 years of age or older

Exclusion Criteria:

* Age <7
* Intercurrent conditions that in the opinion of the investigator would confound the findings of the study.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants with RT-PCR positive for SARS-CoV-2 or diagnosed empirically based on known exposure and symptoms of fever, cough, and shortness of breath. Empirically diagnosed individuals who are negative at baseline by RT-PCR and serology Immunoglobulin M (IgM)/Immunoglobulin G (IgG) will be classified as uninfected and will not participate further, but may be replaced. Negative participants with no known prior COVID-19 diagnosis or COVID-19 vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-03-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Duration of SARS-CoV-2 viral persistence in naso/oropharyngeal samples | Up to 96 weeks
  Duration of SARS-CoV-2 viral persistence defined as the number of days from symptom onset to the most recent positive SARS-CoV-2 PCR naso/oropharyngeal test, as determined by the established cycle threshold cut-off on a validated real-time quantitative reverse transcription polymerase chain reaction (qRT-PCR) assay.
Duration of SARS-CoV-2 viral persistence in stool or rectal swab samples | Up to 96 weeks
  Duration of SARS-CoV-2 viral persistence defined as the number of days from symptom onset to the most recent positive SARS-CoV-2 PCR stool or rectal swab samples, as determined by the established cycle threshold cut-off on a validated qRT-PCR assay.
Duration of SARS-CoV-2 viral persistence in semen samples | Up to 96 weeks
  Duration of SARS-CoV-2 viral persistence defined as the number of days from symptom onset to the most recent positive SARS-CoV-2 PCR semen sample, as determined by the established cycle threshold cut-off on a validated qRT-PCR assay.
Duration of SARS-CoV-2 viral persistence in breast milk samples | Up to 96 weeks
  Duration of SARS-CoV-2 viral persistence defined as the number of days from symptom onset to the most recent positive SARS-CoV-2 PCR breast milk sample, as determined by the established cycle threshold cut-off on a validated qRT-PCR assay.
Prevalence of cell immune responses | Up to 96 Weeks
  Prevalence defined as the number of participants with B cell, cluster of differentiation 4 (CD4), cluster of differentiation 8 (CD8), natural killer (NK), and natural killer T (NKT) cell immune responses. Plasma will be used for evaluation of neutralizing and binding antibody titers to SARS-CoV-2.
Duration of COVID-19 Symptoms | Up to 96 weeks
  The duration, in weeks, of COVID-19 symptoms as assessed by a symptom survey. Participants will complete health surveys at each study visit that include questions regarding COVID-19 symptoms, in addition to general health questions.
Prevalence of post-viral sequelae | Up to 96 weeks
  Prevalence defined as the number of participants that develop post-viral sequelae as assessed by a symptom survey. Participants will complete health surveys at each study visit that include questions regarding COVID-19 symptoms, in addition to general health questions.
Prevalence of SARS-CoV-2 persistence and bacterial/viral community structures | Up to 96 weeks
  Prevalence defined as the number of participants with SARS-CoV-2 persistence and bacterial/viral community structures.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Yin, MD, MS, Principal Investigator — Associate Professor of Medicine
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified patient data, including test results, may be shared with other researchers within Columbia University at the discretion of the Principal Investigator, and only when the Institutional Review Board (IRB) approval has been granted to allow for the sharing of such data.

REFERENCES:
- [Background] Bergantz L, Subra F, Deprez E, Delelis O, Richetta C. Interplay between Intrinsic and Innate Immunity during HIV Infection. Cells. 2019 Aug 17;8(8):922. doi: 10.3390/cells8080922. PMID 31426525
- [Background] 2. New York State Department of Health. https://coronavirus.health.ny.gov/countycounty-breakdown-positive-cases. Accessed March 23, 2020
- [Background] 3. WHO Coronavirus disease 2019, Situation Report-63
- [Background] 4. Discontinuation of Transmission-Based Precautions and Disposition of Patients with COVID-19 in Healthcare Settings (Interim Guidance). https://www.cdc.gov/coronavirus/2019-ncov/hcp/disposition-hospitalized-patients.html. Accessed March 23, 2020.
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Holshue ML, DeBolt C, Lindquist S, Lofy KH, Wiesman J, Bruce H, Spitters C, Ericson K, Wilkerson S, Tural A, Diaz G, Cohn A, Fox L, Patel A, Gerber SI, Kim L, Tong S, Lu X, Lindstrom S, Pallansch MA, Weldon WC, Biggs HM, Uyeki TM, Pillai SK; Washington State 2019-nCoV Case Investigation Team. First Case of 2019 Novel Coronavirus in the United States. N Engl J Med. 2020 Mar 5;382(10):929-936. doi: 10.1056/NEJMoa2001191. Epub 2020 Jan 31. PMID 32004427
- [Background] Severe acute respiratory syndrome (SARS). Wkly Epidemiol Rec. 2003 Mar 21;78(12):81-3. No abstract available. English, French. PMID 12701272
- [Background] Chan KH, Poon LL, Cheng VC, Guan Y, Hung IF, Kong J, Yam LY, Seto WH, Yuen KY, Peiris JS. Detection of SARS coronavirus in patients with suspected SARS. Emerg Infect Dis. 2004 Feb;10(2):294-9. doi: 10.3201/eid1002.030610. PMID 15030700
- [Background] Corman VM, Albarrak AM, Omrani AS, Albarrak MM, Farah ME, Almasri M, Muth D, Sieberg A, Meyer B, Assiri AM, Binger T, Steinhagen K, Lattwein E, Al-Tawfiq J, Muller MA, Drosten C, Memish ZA. Viral Shedding and Antibody Response in 37 Patients With Middle East Respiratory Syndrome Coronavirus Infection. Clin Infect Dis. 2016 Feb 15;62(4):477-483. doi: 10.1093/cid/civ951. Epub 2015 Nov 12. PMID 26565003
- [Background] Haak BW, Littmann ER, Chaubard JL, Pickard AJ, Fontana E, Adhi F, Gyaltshen Y, Ling L, Morjaria SM, Peled JU, van den Brink MR, Geyer AI, Cross JR, Pamer EG, Taur Y. Impact of gut colonization with butyrate-producing microbiota on respiratory viral infection following allo-HCT. Blood. 2018 Jun 28;131(26):2978-2986. doi: 10.1182/blood-2018-01-828996. Epub 2018 Apr 19. PMID 29674425
- [Background] PREVAIL III Study Group; Sneller MC, Reilly C, Badio M, Bishop RJ, Eghrari AO, Moses SJ, Johnson KL, Gayedyu-Dennis D, Hensley LE, Higgs ES, Nath A, Tuznik K, Varughese J, Jensen KS, Dighero-Kemp B, Neaton JD, Lane HC, Fallah MP. A Longitudinal Study of Ebola Sequelae in Liberia. N Engl J Med. 2019 Mar 7;380(10):924-934. doi: 10.1056/NEJMoa1805435. PMID 30855742
- [Background] Kurscheidt FA, Mesquita CSS, Damke GMZF, Damke E, Carvalho ARBA, Suehiro TT, Teixeira JJV, da Silva VRS, Souza RP, Consolaro MEL. Persistence and clinical relevance of Zika virus in the male genital tract. Nat Rev Urol. 2019 Apr;16(4):211-230. doi: 10.1038/s41585-019-0149-7. PMID 30696994
- [Background] Den Boon S, Marston BJ, Nyenswah TG, Jambai A, Barry M, Keita S, Durski K, Senesie SS, Perkins D, Shah A, Green HH, Hamblion EL, Lamunu M, Gasasira A, Mahmoud NO, Djingarey MH, Morgan O, Crozier I, Dye C. Ebola Virus Infection Associated with Transmission from Survivors. Emerg Infect Dis. 2019 Feb;25(2):249-255. doi: 10.3201/eid2502.181011. Epub 2019 Feb 17. PMID 30500321
- [Background] Jacobs M, Rodger A, Bell DJ, Bhagani S, Cropley I, Filipe A, Gifford RJ, Hopkins S, Hughes J, Jabeen F, Johannessen I, Karageorgopoulos D, Lackenby A, Lester R, Liu RS, MacConnachie A, Mahungu T, Martin D, Marshall N, Mepham S, Orton R, Palmarini M, Patel M, Perry C, Peters SE, Porter D, Ritchie D, Ritchie ND, Seaton RA, Sreenu VB, Templeton K, Warren S, Wilkie GS, Zambon M, Gopal R, Thomson EC. Late Ebola virus relapse causing meningoencephalitis: a case report. Lancet. 2016 Jul 30;388(10043):498-503. doi: 10.1016/S0140-6736(16)30386-5. Epub 2016 May 18. PMID 27209148
- [Background] Soka MJ, Choi MJ, Baller A, White S, Rogers E, Purpura LJ, Mahmoud N, Wasunna C, Massaquoi M, Abad N, Kollie J, Dweh S, Bemah PK, Christie A, Ladele V, Subah OC, Pillai S, Mugisha M, Kpaka J, Kowalewski S, German E, Stenger M, Nichol S, Stroher U, Vanderende KE, Zarecki SM, Green HH, Bailey JA, Rollin P, Marston B, Nyenswah TG, Gasasira A, Knust B, Williams D. Prevention of sexual transmission of Ebola in Liberia through a national semen testing and counselling programme for survivors: an analysis of Ebola virus RNA results and behavioural data. Lancet Glob Health. 2016 Oct;4(10):e736-43. doi: 10.1016/S2214-109X(16)30175-9. Epub 2016 Aug 30. PMID 27596037
- [Background] van Doremalen N, Bushmaker T, Morris DH, Holbrook MG, Gamble A, Williamson BN, Tamin A, Harcourt JL, Thornburg NJ, Gerber SI, Lloyd-Smith JO, de Wit E, Munster VJ. Aerosol and Surface Stability of SARS-CoV-2 as Compared with SARS-CoV-1. N Engl J Med. 2020 Apr 16;382(16):1564-1567. doi: 10.1056/NEJMc2004973. Epub 2020 Mar 17. No abstract available. PMID 32182409
- See also: Columbia University Study Link and Eligibility Questionnaire — https://recruit.cumc.columbia.edu/clinical_trial/1940